CLINICAL TRIAL: NCT03053219
Title: An Open-Label, Non-Randomized, Single-Center Study to Preliminary Evaluation of Safety and Efficacy of Patients Who Participant in [14C] AC0010 Trail and Subsequent Receiving AC0010 Treatment
Brief Title: Preliminary Evaluation of Safety and Efficacy by [14C] AC0010 Trail and Subsequent AC0010 Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC201606AVTN07
Record Dates: First submitted 2016-12-19; First posted 2017-02-15 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma，Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC0010 (Experimental): each participant will be given AC0010 300mg bid
  Interventions: Drug: AC0010

INTERVENTIONS:
Drug: AC0010 — Oral dose of 300mg bid,the two doses are advised to be administered at an interval of 12 hours
  Other Names: AC0010MA

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of male Patients With Advanced NSCLC who participant in [14C] AC0010 ADME.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate safety and efficacy of male Patients With Advanced NSCLC who participant in [14C] AC0010 ADME (absorption, distribution, metabolism and excretion) trial and subsequent receiving AC0010 treatment.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* histologically or cytologically confirmed diagnosis of local advanced or recurrent NSCLC
* failed to the treatment of EGFR-TKI and harbored T790M mutation
* male, Age 18~ 65, have a body mass index (BMI)>19 kg/m2
* Eastern Cooperative Oncology Group performance status(ECOG PS):0-1,Life expectancy of more than 3 months
* main organs function is normal, laboratory values as listed below: blood test without blood transfusion within 14 days

  1. Haemoglobin >100 g/L
  2. Absolute neutrophil count ≥2.0x10^9/L or WBC ≥3.5 x10^9/L
  3. Platelet count ≥ 80x10^9/L
  4. Total bilirubin ≤1.5xULN
  5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN)
  6. Serum creatinine ≤1.5xULN or creatinine clearance ratio ≥60 mL/ min
* Any prior treatment (chemotherapy, radiotherapy or surgery) must be completed over 4 weeks(target therapy over 2 weeks) from the screening; Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (CTCAE v 4.03)
* International normalized ratio (INR) ≤ 1.5
* Patients and their partners should be willing to use methods of contraception or total abstinence from start of dosing until 6 months after discontinuing of study treatment
* Patients must withdraw from previous study of [14C] AC0010

Exclusion Criteria:

* Prior treated with AC0010 or allergic to drug or its formulation ingredients
* Patients receiving other anti-tumor therapy
* Impairment of GI disease, renal disorders or liver disease that may significantly alter the absorption and metabolic of AC0010 (e.g., Unable to swallow, liver, kidney or gastrointestinal partial resection, chronic diarrhea and intestinal obstruction)
* HCVAb positive, active hepatitis B (excluding HBV carriers), Hepatitis virus markers positive and receiving anti-virus drugs
* Meningeal metastasis; brain metastasis with whole brain radiotherapy; prior received hormones or mannitol for the brain metastasis
* Previous EGFR-TKI treatment related Interstitial lung disease history
* Known human immunodeficiency virus infection (HIV), other acquired or congenital immunodeficiency disease, or a history of organ transplantation
* Any severe and / or uncontrolled active infections
* Patients receiving concomitant immunosuppressive agents or high-dose corticosteroids
* Any severe and / or uncontrolled medical conditions
* Patients being treated with drugs recognized as being inhibitors or inducers of the liver isoenzyme in the last 4 weeks prior to registration in the current study
* Within 3 days prior to the treatment taking of dragon fruit, pomelo, grapefruit, orange, mango and other fruit may affect drug metabolizing enzymes or juice
* Major surgery, incisional biopsy or traumatic injuries;
* Within 4 weeks prior to the screening patients with bleeding ≥ grade 3, non-healing wound, sever ulcer or bone fracture
* Patients received high dose irradiation treatment or other 14C-labeled drug within 1 year
* Known a history of alcoholism or drug abuse
* Investigator judgment that patient is unsuitable to participate in study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | RECIST tumour assessments every 6 weeks from first dose until objective disease progression, up to approximately 11 months
  To assess the overall Objective Response Rate(ORR) of AC0010 in EGFR T790M mutation-positive patients with advanced NSCLC.

SECONDARY OUTCOMES:
Progression Free Survival | RECIST tumour assessments every 6 weeks from first dose until objective disease progression, up to approximately 11 months
  To assess the Progression Free Survival(PFS) of AC0010 in EGFR T790M mutation-positive patients with advanced NSCLC.
Disease control rate | RECIST tumour assessments every 6 weeks from first dose until objective disease progression, up to approximately 11 months
  To assess the Disease control rate(DCR) of AC0010 in EGFR T790M mutation-positive patients with advanced NSCLC.
Number of adverse events (AE) experienced by patients to assess safety | From date of Signed informed consent forms until 30 days after disease progression, intolerable toxicity or withdrawal from study, approximately up to 18 months)
  To assess the safety of AC0010 in EGFR T790M mutation-positive patients with advanced NSCLC.

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiang Liu, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No